CLINICAL TRIAL: NCT05640245
Title: Phase 2, Randomized, Parallel-group, Double-blind, Placebo-controlled Study of Sonelokimab in Patients With Active Psoriatic Arthritis
Brief Title: Evaluation of Sonelokimab for the Treatment of Patients With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1095-PSA-201
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Arthritis, Psoriatic
Keywords: Arthritis, Psoriatic; Skin Diseases; Joint Diseases; Arthritis; Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Skin Diseases; Joint Diseases; Arthritis; Psoriasis | interventions — sonelokimab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- sonelokimab dose regimen 1 (Experimental): Subjects randomized to this arm will receive assigned sonelokimab dosage regimen 1
  Interventions: Drug: Sonelokimab
- sonelokimab dose regimen 2 (Experimental): Subjects randomized to this arm will receive assigned sonelokimab dosage regimen 2
  Interventions: Drug: Sonelokimab
- sonelokimab dose regimen 3 (Experimental): Subjects randomized to this arm will receive assigned sonelokimab dosage regimen 3
  Interventions: Drug: Sonelokimab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo
  Interventions: Drug: Placebo
- adalimumab (Active Comparator): Subjects randomized to this arm will receive adalimumab
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Sonelokimab — randomized treatment; parallel group
  Other Names: M1095
  Arms: sonelokimab dose regimen 1; sonelokimab dose regimen 2; sonelokimab dose regimen 3
Drug: Placebo — randomized treatment; parallel-group
  Arms: Placebo
Drug: Adalimumab — randomized treatment; parallel-group
  Arms: adalimumab

SUMMARY:
This is a study to demonstrate the clinical efficacy and safety of the nanobody® sonelokimab administered subcutaneously (sc) compared with placebo in the treatment of adult participants with active psoriatic arthritis. The study includes adalimumab treatment as an active reference arm.

DETAILED DESCRIPTION:
Patients will be randomized to receive one of three sonelokimab treatment regimes, adalimumab or placebo. Primary efficacy evaluation will take place at Week 12. Patients will be allocated to a further 12 weeks of treatment with sonelokimab or adalimumab based on response assessment at week 12. In certain countries, treatment will end at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥18 years of age;
2. Participant has a confirmed diagnosis of PsA per the 2006 Classification criteria for Psoriatic Arthritis (CASPAR) with symptoms for ≥6 months prior to the Screening Visit;
3. Participant has active disease (defined by a TJC68 of ≥3 and a SJC66 of ≥3);
4. Participant has either current active PsO or a dermatologist confirmed history of PsO;
5. Participant tests negative for rheumatoid factor (RF) at the Screening Visit;
6. Participant tests negative for anti-cyclic citrullinated peptide (CCP) antibodies at the Screening Visit;
7. Participant must be, in the opinion of the investigator, a suitable candidate for treatment with adalimumab per approved local product information.

Exclusion Criteria:

1. Participant with known hypersensitivity to sonelokimab or any of its excipients;
2. Participant with known hypersensitivity to adalimumab or any of its excipients;
3. Participant who has previously failed on anti-interleukin (IL)-17 therapy;
4. Participant who has previously failed on anti-tumor necrosis factor alpha (TNFα) therapy;
5. Participant who has had previous exposure to more than 2 biologic agents of any type to treat PsA prior to the Screening Visit;
6. Participant who has a diagnosis of chronic inflammatory conditions other than PsO or PsA;
7. Participant who has a diagnosis of arthritis mutilans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Response Rate of participants achieving at least a 50% improvement in the American College of Rheumatology criteria (ACR50) | Week 12
  Proportion of participants who achieve ACR50 compared with baseline

SECONDARY OUTCOMES:
Response Rate of participants achieving at least a 20% improvement in the American College of Rheumatology criteria (ACR20) | Week 2, 4, 8, 12
  Proportion of participants who achieve ACR20 compared with baseline
Psoriasis Area and Severity Index (PASI) 90 | Week 4, 8, 12
  Proportion of participants who achieve PASI90 in the subgroup of participants with psoriasis involving at least 3% body surface area at baseline
Response rate of participants achieving at least a 70% improvement in the American College of Rheumatology criteria | Weeks 2, 4, 8, 12
  Proportion of participants who achieve ACR70 compared with baseline
Leeds Enthesitis Index (LEI) | Weeks 4, 8, 12
  Proportion of participants with resolution of enthesitis (LEI = 0)
Leeds Dactylitis Index (LDI) | Weeks 4, 8, 12
  Change from baseline for Leeds Dactylitis Index
Modified Nail Psoriasis Severity Index (mNAPSI) | Week 12
  Change from baseline for mNAPSI
Psoriasis Area and Severity Index (PASI) 100 | Weeks 4, 8, 12
  Proportion of participants who achieve PASI100 in the subgroup of participants with psoriasis involving at least 3% body surface area at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Reich, M.D., Ph.D. (equ.), Study Director — MoonLake Immunotherapeutics AG
Locations (35):
- United States (2):
  - Clinical Site, Rancho Mirage, California
  - Clinical Site, Duncansville, Pennsylvania
- Bulgaria (6):
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
  - Clinical Site, Varna
- Clinical Site, Ostrava, Czechia
- Estonia (2):
  - Clinical Site, Tallinn
  - Clinical Site, Tartu
- Germany (2):
  - Clinical Site, Hamburg
  - Clinical Site, Herne
- Hungary (4):
  - Clinical Site, Budapest
  - Clinical Site, Szentes
  - Clinical Site, Székesfehérvár
  - Clinical Site, Veszprém
- Poland (14):
  - Clinical Site, Bialystok
  - Clinical Site, Bydgoszcz
  - Clinical Site, Elblag
  - Clinical Site, Gdynia
  - Clinical Site, Krakow
  - Clinical Site, Lodz
  - Clinical Site, Nadarzyn
  - Clinical Site, Nowa Sól
  - Clinical Site, Olsztyn
  - Clinical Site, Poznan
  - Clinical Site, Sochaczew
  - Clinical Site, Swidnica
  - Clinical Site, Warsaw
  - Clinical SIte, Wroclaw
- Spain (4):
  - Clinical Site, Madrid
  - Clinical Site, Sabadell
  - Clinical Site, Santiago de Compostela
  - Clinical Site, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McInnes IB, Coates LC, Mease PJ, Ogdie A, Kavanaugh A, Eder L, Schett G, Kivitz A, McGonagle D, Brennan N, Godwood A, Cullen E, Reich K, Ritchlin CT, Merola JF. Sonelokimab, an IL-17A/IL-17F-inhibiting nanobody for active psoriatic arthritis: a randomized, placebo-controlled phase 2 trial. Nat Med. 2025 Dec;31(12):4160-4171. doi: 10.1038/s41591-025-03971-6. Epub 2025 Oct 6. PMID 41053449